CLINICAL TRIAL: NCT05096442
Title: A Multicenter, Prospective, Randomized, Single-blind, Pivotal Clinical Study to Evaluate the Safety and Efficacy of GENOSS® DCB Versus SeQuent® Please NEO in Patients With Coronary De Novo Lesions
Brief Title: Compare the Safety and Efficacy of Genoss® DCB and SeQuent® Please NEO in Korean Patients With Coronary De Novo Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP-DS1001_DN
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: de novo lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genoss® DCB (Experimental): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: GENOSS® DCB
- SeQuent® Please NEO (Active Comparator): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: SeQuent® Please NEO

INTERVENTIONS:
Device: GENOSS® DCB — Drug Coated Balloon
  Other Names: Paclitaxel Coated PTCA Balloon catheter
  Arms: Genoss® DCB
Device: SeQuent® Please NEO — Drug Coated Balloon
  Other Names: Paclitaxel Coated PTCA Balloon catheter
  Arms: SeQuent® Please NEO

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel Paclitaxel-coated balloon (Genoss® DCB) by demonstrating non-inferiority to in-lesion late lumen loss at 6 months after the procedure in Korean patients with coronary de novo lesions compared with a product of the same category (SeQuent® Please NEO).

DETAILED DESCRIPTION:
In a randomized controlled trial to compare with the same-category drug device (SeQuent® Please NEO), 204 patients with coronary de novo lesions were recruited from a total of 12 institutions, and the enrolled subjects were 1: 1 through randomization.

The ratio was assigned to the test group and the control group, and each of the test or control devices was assigned to receive the procedure.

The primary end point is the in-lesion late lumen loss of the target lesion at 6 months after the procedure, and the secondary end point is the target vessel failure (Composite of cardiac death, TV-MI, and ID-TVR) at 6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years old
* Patients requiring PCI with coronary de novo lesions
* Patients with stable angina pectoris, or unstable angina pectoris, and asymptomatic myocardial ischemia
* Women of childbearing age who agreed to use one or more of the clinically appropriate methods of contraception during the trial period.
* In case of voluntarily deciding to participate in this clinical trial by signing the informed consent form

Inclusion criteria for coronary angiography

* Patients with significant coronary artery stenosis (> 50% diameter stenosis on coronary angiography)
* On coronary angiography, the length of the lesion is less than 34 mm and the diameter of the reference vessel of the coronary artery is 2.0 - 4.0mm.

Exclusion Criteria:

* Patients with ST-segment elevation myocardial infarction (STEMI)
* Patients who are contraindicated in aspirin, heparin, ticagrelor, iopromide, clopidogrel, prasugrel and paclitaxel
* Patients with platelet aggregation or disorders at risk of increased bleeding, such as gastrointestinal ulcers, which limit platelet aggregation inhibitory therapy and anticoagulant therapy
* Patients with a left ventricular ejection fraction of less than 30% on echocardiography
* Patients with renal insufficiency (eGFR<30mL/min)
* Patients with a history of cardiogenic shock
* Pregnant or lactating women
* The patients have a life expectancy of less than 12 months
* Patients who have or currently have medical conditions such as psychiatric disorders that significantly affect this clinical trial
* Patients who, in the investigator's judgment, may not be suitable for this clinical trial or may increase the risk associated with participation in the study
* Patients who are currently participating in other clinical trials or have experience participating in other clinical trials within 90 days from the screening date
* Patients who are unsuitable for the study according to the investigator judges

Exclusion criteria for coronary angiography

* Patients with left main coronary lesion
* Patients with graft vessel lesion
* Patients who cannot apply pre-dilation or fail in pre-dilation to apply medical devices for clinical trials
* Patients with one of the following items after pre-dilation of the target lesion

  * When FFR (Functional measurement) is measured as ≤ 0.8 in large vessels with a reference vessel diameter exceeding 2.75mm (However, depending on the judgment of the investigator, FFR measurement may not be performed.)
  * Patients who need stenting due to vascular dissection that restricts blood flow
  * Residual stenosis > 30%
  * TIMI flow < 3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
in-lesion late lumen loss after percutaneous coronary intervention in patients with coronary de novo lesions | Follow-up angiography at 6 months after the procedure
  late lumen loss between test group and control group evaluated by quantitative coronary analysis in patients with coronary de novo lesions

SECONDARY OUTCOMES:
Restenosis rate after percutaneous coronary intervention in patients with coronary de novo lesions | Follow-up angiography at 6 months after procedure
  Restenosis is defined as a case where the DS(Diameter stenosis) of the reference vessel diameter is 50% or more when the successfully treated lesion is evaluated through coronary angiography.
Target vessel failure(TVF) | at 6 and 12 months after the procedure
  Composite of TVF(cardiac death, TV-MI, and ID-TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Seok Shin, MD, PhD, Principal Investigator — Division of Cardiology, Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

REFERENCES:
- [Derived] Shin ES, Park Y, Lee JY, Her AY, Chon MK, Kim S, Rha SW, Oh GC, Cho DK, Kim B, Bae JW. A Prospective Randomized Trial Comparing 2 Different Paclitaxel-Coated Balloons in De Novo Coronary Artery Disease. JACC Asia. 2025 Jan 7;5(1):15-24. doi: 10.1016/j.jacasi.2024.10.028. eCollection 2025 Jan. PMID 39886190